CLINICAL TRIAL: NCT04007003
Title: An Audit of the Impact of Tailored Information Delivered Via a Digital Learning Platform
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LiMo Audit
Record Dates: First submitted 2019-06-06; First posted 2019-07-05 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- optimal injection technique (Experimental): Subjects will be trained on site regarding optimal insulin injection technique, including avoiding injections in lipohypertrophy areas and proper rotation. Furthermore subjects are provided with access codes to watch online training modules on the Becton Dickinson (BD) and Me(TM) platform
  Interventions: Behavioral: training in optimal insulin injection technique

INTERVENTIONS:
Behavioral: training in optimal insulin injection technique — the training will be delivered in person as well as through online training modules via the BD and Me(TM) platform

SUMMARY:
The study intends to audit the impact of optimal insulin injection technique on clinical parameters and self-care behaviour of insulin treated diabetes patients in a prospective manner with a follow-up of 6 months. The optimal injection technique is delivered through education via a multimodal tailored approach augmented with a digital 'tailorable' patient learning platform .

The study is conducted in multiple sites across Belgium. Diabetes patients with or without lipohypertrophy will be entered into the audit. The end points will include the impact on use of insulin, long term blood glucose control (HbA1c), hypoglycaemia, glucose variability, needle reuse, patient injection habits and clinician education, training and information inputs.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus, or Type 2 Diabetes Mellitus
* Injecting insulin for at least 1 year
* Self-managing injection therapy, including daily glucose monitoring
* Access to a device with internet
* Confident in navigating the internet

Exclusion Criteria:

* Pregnant or likely to become pregnant during study period
* Impaired cognitive ability which would prevent informed consent
* Syringe only user
* Insulin pump user
* Glucagon-Like Peptide (GLP)-1 receptor agonists therapy only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Change in Insulin Use | up to 6 months
  Change in Total Daily Dose of insulin for subjects at baseline and after 6 months; expressed as % and units/24 hrs

SECONDARY OUTCOMES:
Change in Glycemic Control | up to 6 months
  Change in HbA1c for subjects at baseline and after 6 months; expressed as % and mmol/mol
Incidence of Hypoglycemic Events | up to 6 months
  Rate of hypoglycemic events requiring 3rd party assistance in 6 months prior to study start (baseline) and during the 6 months of the study
Change in Needle Re-Use | up to 6 months
  Rate of needle re-use by self-reporting at baseline and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe De Block, MD, Principal Investigator — University Hospital, Antwerp
Locations (9):
- Belgium (9):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Imeldaziekenhuis, Bonheiden
  - Universitair Ziekenhuis Brussel, Brussels
  - UZ Gent, Ghent
  - Virga Jesse Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - AZ Nikolaas, Sint-Niklaas
  - AZ Turnhout, Turnhout
  - AZ Jan Portaels, Vilvoorde

IPD SHARING:
Plan to Share IPD: No